CLINICAL TRIAL: NCT04079361
Title: Non-invasive Prenatal Testing for the Presymptomatic Detection of Pregnancy Complications
Brief Title: Early PrEgnancy Complications Testing
Acronym: ExPECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EC/2019/0056
Record Dates: First submitted 2019-04-01; First posted 2019-09-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pregnancy complication (Other): Intervention: blood samples
  Interventions: Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: Blood samples — Bood samples during prenatal and postnatal visits

SUMMARY:
The aim of this study is the early (presymptomatic) detection of pregnancy complications, which could contribute to a preventive treatment.

DETAILED DESCRIPTION:
Prenatal screening for an early detection of fetal abnormalities and pregnancy related complications is of great importance for both the fetus and the mother. The current follow-up consists of a physical screening (maternal blood pressure, edemas, weight, fundus altitude...), lab screenings (urine culture for screening asymptomatic bladder infection, urine stick for preeclampsia, sugar test for gestational diabetes, measuring cervix length for premature birth, Group B streptococcus screening), ultrasound monitoring (structural inspection, biometrics, placental function ...) and fetal monitoring with cardiotocography.

The recent introduction of the Non-Invasive Prenatal Testing (NIPT) caused a major change in prenatal diagnosis. NIPT allows the early (12 weeks gestational age) detection of chromosomal abnormalities, such as trisomy 21, with a very high sensitivity and specificity.

Trisomy 21 is with its incidence of 1/1000 live births only the tip of the iceberg of many other fetal abnormalities and gestational complications that can occur. Pregnancy complications, such as pre-eclampsia, intra-uterine growth retardation (IUGR) and preterm birth have a much higher incidence (up to 5-8% of all pregnancies) and are an important cause of maternal and neonatal morbidity and mortality.

The aim of this study is the early (presymptomatic) detection of pregnancy complications, which could contribute to a preventive treatment. Studies have shown that the major cause of these complications originate from defects in spiral artery remodeling and trophoblast invasion or an abnormal functioning placenta, during the 1st or 2nd trimester. Insufficient oxygen and nutrient flow to the placenta, caused by abnormal (narrowed diameter) spiral arteria, is the most proven underlying origin. These obstructing conditions can lead to a placenta in stress (hypoxia), and therefore potentially a fetus in stress (IUGR). General known is that these pathologies will lead to a different gene expression, which can be investigated by direct analysis of placental RNA (transcriptome) and DNA (methylation profiling). During the last decade, several high impact researchers (for example the research groups of Dennis Lo and Stephen Quake, founders of the current worldwide NIPT screening) have investigated gene expression profiles in the placenta in normal and complicated pregnancies, by analyzing the placental cell free DNA and RNA present in maternal plasma. Very recent findings indicate a huge potential in non-invasively profiling the placental transcriptome and methylome. Advances in next-generation sequencing and molecular analysis made it possible to measure circulating nucleic acids to improve the investigator's understanding of placental pathology and develop novel non-invasive biomarkers for pregnancy complications and monitoring high-risk pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Every pregnant woman, speaking and understanding Dutch, French or English

Exclusion Criteria:

* not able to understand and adhere to the informed consent and study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Optimizing and validating a non-invasive prenatal genetic screening for the early presymptomatic detection of pregnancy complications | Through study completion, an average of 30 weeks
  The placental transcriptome represents gene expression in this specific tissue. Abnormalities in the placenta have been shown to lead to aberrant gene expression patterns. The RNA biomarker (transcript) analysis will be performed by RNA sequencing of cell free RNA by next generation sequencing. After sequencing, RNA molecules will be identified and transcripts will be quantified and evaluated between normal and pregnancies with complications. This will provide information regarding aberrant expressed genes and transcripts. Statistical analysis between both groups will be performed to identify and subsequently validate biomarkers that can be used to presymptomatically prediction pregnancy complications.
Optimizing and validating a non-invasive prenatal genetic screening for the early presymptomatic detection of pregnancy complications | Through study completion, an average of 30 weeks
  Epigenetic modifications (eg. DNA methylation) can alter gene expression, without altering the DNA sequence itself. DNA methylation can be investigated by bisulfite conversion of the DNA followed by next-generation sequencing. It has been shown that complicated pregnancies have aberrant methylation profiles of placental DNA. By analyzing the methylation profile of the cell free DNA of normal and complicated pregnancies and performing a statistical analysis, we will identify biomarkers and set-up a prediction model for the prediction of pregnancy complication.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Dehaene, MD, Principal Investigator — UZ Gent
Locations (1):
- Ghent University Hospital - Women's Clinic, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided